CLINICAL TRIAL: NCT02508142
Title: Assessment of Analgesic Efficacy and Safety of Intravenous Hyoscine-N-Butylbromide in Patients With Abdominal Colic Associated With Acute Gastroenteritis; a Randomized, Double-blind, Placebo Controlled Study
Brief Title: Analgesic Efficacy of Intravenous Hyoscine-N-Butylbromide (HNB) in Abdominal Colic Associated With Acute Gastroenteritis
Acronym: HNB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Elif Yaka, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KocaeliU
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Abdominal Cramps
MeSH Terms: conditions — Colic | interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyoscine-N-Butylbromide (Active Comparator): 20 mg Hyoscine-N-Butylbromide in 98 mL normal saline (totally 100 mL)
  Interventions: Drug: Hyoscine-N-Butylbromide
- Placebo (Placebo Comparator): 100 mL normal saline
  Interventions: Drug: Hyoscine-N-Butylbromide

INTERVENTIONS:
Drug: Hyoscine-N-Butylbromide — Study Drug: 20 mg/2 mL Hyoscine-N-Butylbromide in 98 mL normal saline (totally 100 mL) ıntravenous form of Hyoscine-N-Butylbromide in normal saline is in the same appearance with placebo Study drug: 100 mL normal saline (placebo) (totally 100 mL)
  Drug: Fentanyl 1 mcg/kg as rescue analgesia at 30th minute
  Other Names: Buscopan, 20mg/2 mL (Boehringer Ingelheim İlaç Ticaret A.Ş)

SUMMARY:
This study aims to assess the analgesic efficacy and safety of intravenous 20 mg Hyoscine-N-Butylbromide versus placebo for the treatment of abdominal colic associated with acute gastroenteritis in the emergency department.

DETAILED DESCRIPTION:
Acute gastroenteritis is a frequent cause of emergency department (ED) presentation. Mainstays of ED treatment are rehydration and antiemetics when needed. Since crampy abdominal pain accompanies (diarrhea) acute gastroenteritis in 67-90% of patients, emergency physicians may have to deal with spasmodic colics in these patients.

Hyoscine-N-butylbromide (HNB), is an anticholinergic agent which has been in use as an antispasmodic agent for sixty years all over the world. It has been studied and revealed various efficacy for several conditions (e.g; biliary colic, renal colic, endoscopic interventions, radiologic interventions, during labor, nonspecific abdominal pain and irritable bowel syndrome).

HNB is commonly used for symptomatic relief of abdominal cramps associated with acute gastroenteritis in the EDs, whereas the literature lacks evidence regarding its efficacy and safety for this condition.

The aim of this study is to assess the analgesic efficacy and safety of intravenous 20 mg hyoscine-n-butylbromide versus placebo in patients with abdominal colic associated with acute gastroenteritis in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Presenting to the emergency department with abdominal cramps associated with acute gastroenteritis
* The pain intensity score upon screening is at least 20 mm on visual analog scale
* Patients who agree to participate and sign the informed consent

Exclusion Criteria:

* Patients younger than 18 years
* Pain of > 7 days
* Use of any analgesic within 6 hours of ED presentation
* Concomitant medication with spasmolytics, anticholinergics, drugs affecting gastrointestinal motility such as metoclopramide, loperamide, opioid analgesics
* Patients who were administered dopamine antagonists before screening
* Documented or self-reported hypersensitivity to hyoscine-n-butylbromide
* Confirmed or suspected pregnancy
* Breastfeeding
* Glaucoma
* Myasthenia gravis
* Benign prostatic hyperplasia or urinary obstruction
* Any suspected other cause of acute abdominal pain
* Peritonism
* Mechanical stenosis of the gastrointestinal tract, paralytic ileus, megacolon
* Previous intestinal resection
* History of inflammatory bowel disease
* Tachyarrhythmia
* Severe dehydration requiring fluid resuscitation immediately
* Unable to consent
* Refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in the mean pain intensity scores on visual analog scale | 15, 30, 60 minutes
  Change in the mean pain intensity scores on visual analog scale

SECONDARY OUTCOMES:
Adverse events | 6 hours
  any adverse reactions
Incidence of rescue analgesia | at 30 minute
  Incidence of rescue analgesia (Fentanyl 1mcg/kg) requirement

CONTACTS AND LOCATIONS:
Overall Officials: Elif YAKA, M.D., Principal Investigator — Kocaeli University, Faculty of Medicine, Emergency Department
Locations (1):
- Kocaeli University, Faculty of Medicine, Emergency Departmentt, Kocaeli, Turkey (Türkiye)